CLINICAL TRIAL: NCT00813813
Title: Phase I/II, Multicenter, Open-label, Single Administration, Dose Finding, Clinical Trial to Evaluate the Safety and Tolerability of Intradiscal rhGDF-5 for the Treatment of Early Stage Lumbar Disc Degeneration
Brief Title: Intradiscal rhGDF-5 Phase I/II Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-Intradiscal rhGDF-5-01
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-01

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intradiscal rhGDF-5 (Experimental): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.
  Interventions: Drug: Intradiscal rhGDF-5

INTERVENTIONS:
Drug: Intradiscal rhGDF-5 — The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic protein (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc. In vitro experiments have shown that rhGDF-5 can stimulate gene expression and synthesis of the extracellular matrix proteins type II collagen and aggrecan. In vivo experiments in rabbit models of disc degeneration have shown that intradiscal injections of rhGDF-5 can stimulate an increase in disc height and hydration.

SUMMARY:
Study to show the effectiveness and safety of a single injection of rhGDF5 into a degenerating single spinal disc in treating lumbar level degenerative disc disease

ELIGIBILITY:
Inclusion Criteria:

1. Persistent low back pain, with at least 3 months of non-surgical therapy, at one symptomatic lumbar level (L3/L4 to L5/S1) as confirmed using a standardized discography protocol
2. Oswestry Disability Index of 30 or greater
3. Low back pain score greater than or equal to 4 cm as measured by VAS, at Visit 1 baseline and on day of treatment to confirm eligibility prior to administration

Exclusion Criteria:

1. Persons unable to have a discogram, CT or an MRI
2. Abnormal neurological exam at baseline (e.g., radiculopathy)
3. Radicular pain
4. Leak of contrast agent during the discogram, into the epidural space (does not include leak of contrast agent along the needle track)
5. MRI findings demonstrate any of the following:· Suspected disc appears normal· >50% decrease in disc height· Modic changes, and/or· Presence of osteophytes or significant facet arthrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Rathmell, MD, Principal Investigator — Massachusetts General Hospital; Richard Guyer, MD, Principal Investigator — Texas Back Institute; Marvin Tark, MD, Principal Investigator — Drug Study America; Jim Youssef, MD, Principal Investigator — Durango Orthopedic Associates/Spine Colorado; Norman Harden, MD, Principal Investigator — Shirley Ryan AbilityLab; Jonathan Borden, MD, Principal Investigator — Riverhills Healthcare, Inc.; Yaoming Gu, MD, Principal Investigator — Virginia Commonwealth University
Locations (8):
- United States (8):
  - Spine Institute, Santa Monica, California
  - Durango Orthopedic Associates/Spine Colorado, Durango, Colorado
  - Drug Studies America, Marietta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Riverhills Healthcare, Inc., Cincinnati, Ohio
  - TBI Clinical Research, LLC, Plano, Texas
  - Virginia Commonwealth University Spine Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Intradiscal rhGDF-5 (0.25mg); Intradiscal rhGDF-5 (1.0mg): The API is recombinant human growth and differentiation factor-5 (rhGDF-5), a recombinant version of human GDF-5. GDF-5 is a member of the transforming growth factor-b (TGF-b) superfamily and the bone morphogenetic (BMP) subfamily, and is known to influence the growth and differentiation of various tissues, including the intervertebral disc.
Period: Overall Study
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Started | 7 | 25
Completed | 4 | 16
Not Completed | 3 | 9
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 7
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg) | Total
Number analyzed (Participants) | 7 | 25 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (5.92) | 44.4 (8.63) | 41.7 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 1 | 12 | 13
Region of Enrollment [Number; unit: participants]
  United States | 7 | 25 | 32

OUTCOME MEASURES:

1. Primary Outcome: Neurological Assessment for Motor Function and Reflexes/Sensory
Description: Neurological Assessment for Motor Function and Reflexes/Sensory- Number of patients with Clinically Significant Abnormal results at 12 months.
  For Motor Function, Clinically Significant Abnormal results are determined by the surgeon investigator and are further classified by grade: 0= No Movement, 1= Flicker/trace of contraction, 2=Active movement when gravity removed, 3= Active movement against gravity, 4= Active Movement against gravity and resistance.
  For Reflexes/Sensory, Clinically Significant Abnormal results are determined by the surgeon investigator and are based on exams of the Knee, Ankle, L3-L5 Dermatone, and S1 Dermatome. Tension signs are evaluated with a straight leg raise to determine at which point, if any, sciatic pain occurs.
Time Frame: 12 months
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
participants | 0 | 0

2. Secondary Outcome: Change in Function Assessed by Oswestry Disability Index Change at 12 Months From Baseline
Description: The Oswestry Disability Index (ODI) is a 10-category (Pain Intensity, Personal Care, Lifting, Walking, Sitting, Standing, Sleeping, Sex Life, Social Life, Traveling) disability measurement scale with a graded response from 0 to 5, with 0 being the best score (no impairment) to 5 being the worst score (significant impairment). ODI score for a subject is calculated by adding the scores and converting the score to a 100 point scale.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
units on a scale | -10.0 (12.00) | -17.0 (18.00)

3. Primary Outcome: Treatment Emergent Adverse Events- Relationship to Study Drug
Description: Number of patients with Treatment Emergent Adverse Events that were designated as related or possibly related to Study Drug.
Time Frame: Through a 12 month period and annual telephone contact at 24 and 36 months for subject health status follow-up
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
participants | 2 | 1

4. Secondary Outcome: Change in Pain Visual Analog Scale (VAS) at 12 Months From Baseline
Description: The Visual Analog Scale (VAS) pain score asks the subject to place a vertical mark on a horizontal line (that is approximately 10 cm long) with 'No Pain' (score of 0 = 0 cm) listed on the left and 'Very severe pain' (score of 10=10cm) labeled on the right. The subject is instructed to indicate the amount of pain they feel in their back.
Time Frame: 12 months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
units on a scale | -2.0 (2.00) | -3.0 (2.00)

5. Secondary Outcome: Change in Physical Component Summary of Quality of Life Measure Assessed by Short-Form 36 at 12 Months From Baseline
Description: The 36-item Short Form Health Survey (SF-36) is a patient reported outcome survey that evaluates functional health and well-being. The survey is converted into two summary measures (the Physical Component - PCS and Mental Component- MCS) that are scored from 0 to 100 (where 100 indicates the highest level of health).
Time Frame: 12 Months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
units on a scale | 5.0 (6.00) | 8.0 (10.00)

6. Secondary Outcome: Change in Mental Component Summary Quality of Life Measure Assessed by Short Form SF-36 at 12 Months From Baseline
Description: as for outcome 5
Time Frame: 12 Months
Population: FAS Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Number analyzed (Participants) | 7 | 25
units on a scale | 7.0 (8.00) | 3 (12.00)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through a 12 month period and annual telephone contact at 24 months and 36 months
Arm/Group | Intradiscal rhGDF-5 (0.25mg) | Intradiscal rhGDF-5 (1.0mg)
Serious Adverse Events (participants affected / at risk) | 2/7 | 2/25
Other Adverse Events (participants affected / at risk) | 7/7 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (0.25mg) (N=7) | Intradiscal rhGDF-5 (1.0mg) (N=25)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intradiscal rhGDF-5 (0.25mg) (N=7) | Intradiscal rhGDF-5 (1.0mg) (N=25)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 14 (16)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint Instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Accidental Needle Stick (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 5 (6)
Injection Site Bruising (General disorders) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Mood Swings (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Ovarian Mass (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (2) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Investigators may freely present or publish results of the Clinical Investigation in a manner which fairly sets forth the conclusions reached by the Clinical Investigators, but only after the Sponsor has been given the opportunity of reviewing the proposed presentation or publication at least 60 days prior to the intended submission, presentation, or publication date.